CLINICAL TRIAL: NCT03399292
Title: Effect of Lipid Based Eye Drops on Tear Film Lipid Layer Thickness in Subjects With Dry Eye Disease, Meibomian Gland Dysfunction, Blepharospasm and Healthy Subjects - a Pilot Study
Brief Title: Effect of Lipid Based Eye Drops on Tear Film Lipid Layer Thickness
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc.Prof.PD MD, Medical University of Vienna
Other Study IDs: OPHT-031116
Record Dates: First submitted 2018-01-08; First posted 2018-01-16 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2022-04

CONDITIONS: Dry Eye Syndromes
Keywords: Lipid based eye drops; Tearfilm lipid layer thickness
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Group 1: 10 male and female healthy subjects receive Cationorm MD sine eye drops once
  Interventions: Drug: Cationorm MD sine eye drops
- Group 2: 10 male and female volunteers with dry eye disease receive Cationorm MD sine eye drops once
  Interventions: Drug: Cationorm MD sine eye drops
- Group 3: 10 male and female volunteers with Maibomian gland disease receive Cationorm MD sine eye drops once
  Interventions: Drug: Cationorm MD sine eye drops
- Group 4: 10 male and female volunteers with receive Cationorm MD sine eye drops once
  Interventions: Drug: Cationorm MD sine eye drops

INTERVENTIONS:
Drug: Cationorm MD sine eye drops — studyparticipants receive lipidbased eye drops once only in the study eye

SUMMARY:
Dry eye disease (DED) is a common ocular disease, especially in the elderly population. Despite many treatment approaches, instillation of topical lubricants remains the mainstay of therapy. However, most of the topical lubricants available are not very well characterised and data about efficacy is sparse.

The aim of the present pilot study is to investigate the effect of topically administered lipid based eye drops on tear film lipid layer thickness in subjects with dry eye disease, Meibomian gland dysfunction, blepharospasm and healthy subjects.

Tear film lipid layer and tear film thickness will be assessed using the Lipiview II interferometer and OCT. Measurements will be performed before instillation of the eye drops and every 10 minutes after instillation for one hour. One eye will receive lipid based eye drops, the other eye will receive no eye drops and will be used as control. The study eye will be chosen randomly. In addition, Dynamic Meibomian gland imaging, Schirmer I test, corneal fluorescein staining and determination of tear break up time (BUT) will be performed

ELIGIBILITY:
Inclusion Criteria:

All groups

* Men and women aged over 18 years
* Normal findings in the medical history unless the investigator considers an abnormality to be clinically irrelevant
* Ametropy < 6 dpt
* No application of eye drops or ointments in the 24 hours preceding the screening visit as well as the study day Dry eye disease group
* History of dry eye disease ≥ 3 months
* Schirmer I test ≤ 10 mm and ≥ 2 mm or BUT ≤ 10 sec
* Normal ophthalmic findings with the exception of DED Meibomian gland disease group
* Dry eye disease most likely caused by MGD, no other cause identifiable which is more likely (e.g. intake of concomitant medication that could induce DED, systemic diseases such as systemic arthritis or diabetes), as judged by the investigator
* History of dry eye disease ≥ 3 months
* Normal ophthalmic findings except dry eye disease
* BUT ≤ 10 seconds Blepharospasm group
* Clinical diagnosis of blepharospasm
* Normal ophthalmic findings with the exception of blepharospasm and dry eye
* Schirmer I test > 10 mm and BUT > 10 sec

Exclusion Criteria:

All groups

* Clinically relevant illness in the 3 weeks before the screening or study day
* Ametropy ≥ 6 dpt
* Pregnancy or planned pregnancy
* Difference of more than 5 mm in Schirmer I test or difference of > 3 sec in BUT between the two eyes
* Known medical history of allergy, hypersensitivity or poor tolerance to any components of the medical device used in the study
* Treatment with topical or systemic steroids, immune suppressants, NSAIDs: ongoing or in the last 4 weeks
* Treatment with medication known to have a detrimental effect on tear film (e.g. antidepressants, anxiolytics, neuroleptics, antihistaminic drugs, cholinergic drugs, antimuscarinic drugs, phenothiazine, beta blockers): treatment duration ≤ 4 weeks or changed dose since ≤ 4 weeks or during the study
* Alcohol abuse
* Contact lens wear Meibomian gland dysfunction group
* Sjögren's syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10 healthy male and female volunteers 10 male and female subjects with dry eye disease 10 male and female subjects with Meibomian gland dysfunction 10 male and female subjects with blepharospasm
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2024-11-26 (Actual)

PRIMARY OUTCOMES:
Tear film lipid layer thickness as measured with Lipiview II | 12.04.2017-30.12.2018

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No